CLINICAL TRIAL: NCT07286331
Title: A Randomized, Open-label, Multicenter, Phase 3 Study to Investigate GSK5733584 Compared With Chemotherapy in Participants With Recurrent Endometrial Cancer
Brief Title: A Study to Investigate GSK5733584 Compared With Chemotherapy in Participants With Recurrent Endometrial Cancer (BEHOLD-Endometrial01)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 224038; 2025-523362-25-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-12; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Neoplasms, Endometrial
Keywords: Endometrial Cancer; GSK5733584; Paclitaxel; Doxorubicin; Antibody-drug conjugate; BEHOLD-Endometrial01
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Paclitaxel; Doxorubicin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The independent central reviewer assessing primary outcome data will be masked (blinded) from participants treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK5733584 (Experimental): Participants will receive GSK5733584
  Interventions: Drug: GSK5733584
- Standard of Care (Active Comparator): Participants will receive standard of care treatment (Paclitaxel or Doxorubicin) as per investigator's discretion
  Interventions: Drug: Paclitaxel; Drug: Doxorubicin

INTERVENTIONS:
Drug: GSK5733584 — GSK5733584 will be administered
  Arms: GSK5733584
Drug: Paclitaxel — Paclitaxel will be administered
  Arms: Standard of Care
Drug: Doxorubicin — Doxorubicin will be administered
  Arms: Standard of Care

SUMMARY:
This study specifically aims to evaluate how well GSK5733584 works in treating Endometrial Cancer (EC) compared to standard of care. The study also assesses whether GSK5733584 is safe and tolerated well by participants in comparison to standard of care and will help provide a better understanding of the main side effects of the drugs

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Is at least 18 years of age and the legal age of consent in the jurisdiction in which the study is taking place at the time of signing the Informed consent form (ICF).
* Has histologically confirmed recurrent or persistent endometrial carcinoma including but not limited to endometroid, serous, clear cell, and endometrial carcinosarcoma. Mixed epithelial carcinomas are permitted.
* Has undergone at least 1 and no more than 2 lines of prior systemic treatment for EC. Up to 3 lines of prior systemic treatment are acceptable if one line was administered in the adjuvant/neo-adjuvant setting. The definition of prior lines of therapy is as follows:

  * Adjuvant ± neo-adjuvant therapy counts as one line of treatment.
  * Maintenance therapy is considered part of the preceding line and does not count as an independent line.
  * Switching to another agent within the same class due to toxicity (without disease progression) is considered part of the same line of therapy.
  * Unplanned addition or switching to a new drug in a different class is considered a separate line of therapy.
  * Hormonal therapy is NOT counted as a separate line.
* Must have received prior platinum-based chemotherapy and anti- Programmed cell death 1 (PD-1) /anti- Programmed cell death ligand 1 (PD-L1) therapy, either separately or in combination. Participants deemed unsuitable for a prior PD-1/PD-L1 inhibitor therapy (contraindications such as immunodeficiency, autoimmune disease that required systemic treatment) as determined by the investigator or treating physician are eligible.
* Participants must have a platinum-free interval of less than 12 months if they previously received platinum-based therapy solely in the adjuvant setting.

  * If PD-L1/PD-1 inhibitor therapy was administered with platinum-based treatment, participant is eligible regardless of whether the Platinum-free interval (PFI) exceeds 12 months.
  * Participants with metastatic disease who underwent treatment including gynecological surgery followed by a platinum-based regimen, or those deemed intolerant to platinum-based therapy, are eligible regardless of whether the PFI exceeds 12 months.
* Has provided a Formalin-fixed, paraffin-embedded (FFPE) tumor tissue sample sufficient for the central assessment of B7 homolog 4 protein (B7-H4) expression, with the result of B7-H4 expression testing available prior to date of randomization.
* Has ≥1 Target Lesion per RECIST 1.1 by BICR eligibility review of screening scans.
* Is willing to use adequate contraception. Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and 1 of the following conditions applies:

  * Is a Participant of non-childbearing potential (PONCBP) OR
  * Is a Participant of childbearing potential (POCBP) and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, 30 days prior to Cycle 1 Day 1 (C1D1) and during the study intervention period and for at least 8 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first dose of study intervention.
* A POCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention

  * If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
  * Additional requirements for pregnancy testing during and after study intervention are described in protocol.
  * The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a participant with an early undetected pregnancy.
* Is capable of giving signed informed consent including compliance with the requirements and restrictions listed in the ICF and in the protocol.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has adequate organ function.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Mesenchymal tumors of the uterus (uterine sarcomas) and neuroendocrine uterine cancer.
* Has a malignancy (except disease under study) that has progressed or required active treatment within the past 36 months prior to date of randomization except for basal cell or squamous cell carcinomas of the skin or in-situ carcinomas [e.g., breast, cervix, bladder] that have been resected with no evidence of metastatic disease, or that is otherwise considered cured by the investigator.
* Has any history of prior allogenic or autologous bone marrow transplant or other solid organ transplant.
* Has known sensitivity to study intervention components or excipients or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Has untreated brain or Central nervous system (CNS) metastases or brain/CNS metastases that have progressed (e.g., evidence of new or enlarging brain metastasis or new neurologic symptoms attributable to brain/CNS metastases). Participants with previously treated and clinically stable brain/CNS metastases and who have completed all corticosteroid therapy for ≥14 days before date of C1D1 are not excluded from participation.
* Has any evidence of current Interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or non-infectious pneumonitis.
* Has ongoing adverse reaction(s) from prior therapy that has (have) not recovered to ≤ Grade 1 or to the baseline status preceding prior therapy, excluding alopecia, hearing loss, vitiligo and endocrinopathy managed with replacement therapy, or that the investigator, with the agreement of the sponsor, considers to be stable or not clinically relevant for the tolerability of study intervention in the current clinical study.
* Has any serious and/or unstable medical or psychiatric disorder or other condition(s) (including laboratory assessment abnormalities) that could interfere with the participant's safety, obtainment of informed consent, or compliance to the study procedures.
* Has had any major surgery within 28 days prior to date of C1D1 or history of local radiotherapy within 21 days prior to C1D1.
* Has received treatment with an investigational agent within 30 days prior to C1D1.
* Has received prior therapy with Topo1i (e.g. irinotecan or topotecan) or ADC with a Topo1i warhead, or B7-H4 targeted therapy.
* Has received treatment with any cytotoxic chemotherapy drugs or other antitumor drugs (including endocrine therapy, molecular targeted therapy, immunotherapy, biotherapy and investigational drug) within 30 days or 5 half-lives, whichever is shorter, prior to C1D1; or need to continue these drugs during the study.
* Has received any live vaccine within 30 days prior to C1D1.Note: mRNA and adenoviral-based Coronavirus disease 2019 (COVID-19) vaccines are considered non-live.
* Has received treatment with strong or moderate inhibitor of Cytochrome P450 (CYP) 3A4 or CYP2D6, strong or moderate inducer of CYP3A, inhibitor of P-glycoprotein (P-gp) or Breast cancer resistant protein (BCRP), or inducer of P-gp within 14 days prior to date of C1D1 or anticipates their use during study participation and up to 30 days after last dose of study intervention.
* Has used drugs known to prolong the QT interval or potentially cause torsades de pointes; or need to continue these medications during the study
* Has received any transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including Granulocyte colony stimulating factor (G-CSF), Granulocyte-macrophage colony stimulating factor (GM-CSF), or recombinant erythropoietin) within 14 days prior to C1D1.
* Has a known Human immunodeficiency virus (HIV) infection AND meets at least 1 of the following criteria:

  * Has documented evidence of plasma HIV-1 Ribonucleic acid (RNA) ≥50 c/mL within 3 months prior to or at screening. In the 3 to 12 months prior to screening, plasma HIV1 RNA levels consistently <50 c/mL are required for enrollment; if multiple instances of plasma HIV-1 RNA values ≥50 c/mL occurred in the 3 to 12 months prior to screening, the participant is not eligible for enrollment unless, per the investigator's assessment, the elevations were neither persistent nor associated with antiretroviral resistance; OR
  * Has not had Cluster of differentiation (CD)4 cell counts measured in the past 12 months (i.e., at least 2 separate measurements taken a minimum of 28 days apart, 1 of which must be conducted at screening); OR
  * Has had any CD4 cell count values ≤350 cells/mm3 in the past 12 months; OR
  * Has had 1 or more changes in their combination antiretroviral therapy regimen or has received an antiretroviral therapy regimen that is inconsistent with locally recommended guidelines during the 3 months prior to screening; OR
  * Has a history of HIV-associated non-Hodgkin lymphoma within 5 years prior to screening or a history of HIV-associated invasive cervical cancer; OR
  * Has received treatment with an HIV1 immunotherapeutic vaccine within 90 days prior to screening.
* Has an Alanine aminotransferase (ALT) value >2.5× Upper limit of normal (ULN) and/or for participants documented liver metastases/tumor infiltration has an ALT value >5x ULN
* Has a total bilirubin value >1.5x ULN.
* Has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, or persistent jaundice.
* Has documented presence of Hepatitis B surface antigen (HBsAg) and/or Hepatitis B core antibody (HBcAb) at screening unless they meet both the following criteria:

  * Participants with chronic Hepatitis B virus (HBV) infection (HBsAg+) or positive HBcAb are required to be receiving effective antiviral therapy (i.e., with nucleos(t)ide analogs [Tenofovir or Entecavir]) for at least 14 days prior to C1D1 and are willing to continue for at least 6 months after treatment discontinuation or longer at the discretion of the treating hepatologist.
  * HBV Deoxyribonucleic acid (DNA) must be adequately suppressed, as per institutional or local guidelines, prior to initiation of study intervention.
* Has a positive Hepatitis C virus (HCV) antibody test result at screening or within 3 months prior to C1D1 unless HCV RNA is negative, indicating past resolved HCV infection, including participants who have undergone curative treatment.
* Has a positive HCV RNA test result at screening or within 3 months prior to C1D1.
* Has QTc >470 milliseconds (msec)
* Has a history of congenital long QT syndrome or a history within 12 months prior to screening of clinically significant or uncontrolled cardiac disease, acute myocardial infarction, New York Heart Association Class III or IV congestive heart failure [NYHA 1994], or clinically significant arrhythmia not controlled by standard of care therapy.
* Participants receiving Doxorubicin ONLY: Has baseline Left ventricular ejection fraction (LVEF) <50% or less than institutional lower limit of normal.
* Has any active renal condition (e.g., infection, requirement for dialysis, or any other significant renal condition that could affect the participant's safety).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2026-03-05 (Estimated); Primary Completion 2028-01-19 (Estimated); Study Completion 2029-03-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by BICR | Up to approximately 97 weeks
  ORR is defined as the percentage of participants with best overall confirmed response of either complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) by Blinded independent central review (BICR)
Progression Free Survival (PFS) by BICR | Up to approximately 97 weeks
  PFS is defined as the time from the date of randomization to the date of first documented Progressive Disease (PD) or death from any cause, whichever occurs first per RECIST 1.1 by BICR assessment

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 156 weeks
  OS is defined as the time from the date of randomization to the date of death due to any cause
ORR by investigator assessment | Up to approximately 156 weeks
  ORR is defined as the percentage of participants with best overall confirmed response of either CR or PR per RECIST 1.1 by investigator assessment
Duration of Response (DOR) by BICR | Up to approximately 156 weeks
  DOR is defined as the time from the date of the first documented objective response (CR or PR) that is subsequently confirmed to the date of first documented PD or death due to any cause, whichever occurs first per RECIST 1.1 by BICR assessment
DOR by investigator assessment | Up to approximately 156 weeks
  DOR is defined as the time from the date of first documented objective response (CR or PR) that is subsequently confirmed to the date of first documented PD or death due to any cause, whichever occurs first per RECIST 1.1 by investigator assessment
PFS by investigator assessment | Up to approximately 156 weeks
  PFS is defined as the time from the date of randomization to the date of first documented PD or death due to any cause, whichever occurs first per RECIST 1.1 by investigator assessment
Number of participants with Treatment-emergent adverse event (TEAEs), Adverse event of special interest (AESIs) and Treatment-emergent serious adverse event (TESAEs) | Up to approximately 156 weeks
Number of participants with TEAEs/AESIs/TESAEs leading to dose modifications or study intervention discontinuation | Up to approximately 156 weeks
Number of participants with changes in vital signs, laboratory tests (hematology and clinical chemistry), and Electrocardiogram (ECG) | Up to approximately 156 weeks
Change from baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) score | Up to approximately 156 weeks
  The EORTC QLQ-C30 includes 30-item questionnaire for evaluating the health-related quality of life (HRQoL) of endometrial cancer participants. These include functional scales, symptom scales, global health status scale, and single item scales. Scores are averaged and transformed to 0 to 100. Higher scores indicate greater functioning, better global health status, or more severe symptoms
Change from baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Endometrial Cancer Module 24 (EORTC QLQ-EN24) | Up to approximately 156 weeks
  The EORTC QLQ-EN24 is a 24-item questionnaire designed as a supplement to the EORTC QLQ-C30 for evaluating quality of life of endometrial cancer participants. Scores are averaged and transformed to a 0 to 100 scale. Higher scores indicate more severe symptoms.
Time to deterioration (TTD) of EORTC QLQ-EN24 | Up to approximately 156 weeks
  TTD is defined as the time from date of randomization to the date of first confirmed clinically meaningful deterioration on any of the following domains: lymphedema, urological symptoms, gastrointestinal symptoms, and pain in back and pelvis domains
TTD of EORTC QLQ-C30 | Up to approximately 156 weeks
  TTD is defined as the time from date of randomization to the date of first confirmed clinically meaningful deterioration on any of the following domains: Physical Functioning, Role Functioning, and Global Health Status/QoL
Number of participants with severity and/or interference of symptomatic AEs as assessed by patient-reported outcome Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to approximately 156 weeks
  The PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicities in participants in cancer clinical trials. The PRO-CTCAE includes an item library of 124 items representing 78 symptomatic toxicities drawn from the CTCAE.
Serum concentration of GSK5733584 (conjugated antibody and payload) | Up to approximately 156 weeks
Number of participants with Antidrug antibody (ADA) and Neutralizing Antibody (NAb) against GSK5733584 | Up to approximately 156 weeks
Titers of ADA against GSK5733584 | Up to approximately 156 weeks

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf